CLINICAL TRIAL: NCT02404584
Title: The Pharmacokinetic Variability of Sunitinib in Patients With Metastatic Renal Cancer: Searching for Pharmacogenetic Determinants
Brief Title: The Pharmacokinetic Variability of Sunitinib in Patients With Metastatic Renal Cancer
Acronym: GenCInibs-Suni
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2014/LM-01bis; 2014-005534-55 (EudraCT Number)
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Kidney Neoplasms
Keywords: Metastatic kidney cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: Patients with kidney cancer and will be starting treatment via sunitinib at the study start will be included.
  Intervention: Blood drawn for genotyping Intervention: Blood drawn for pharmacokinetic measures
  Interventions: Genetic: Blood drawn for genotyping; Biological: Blood drawn for pharmacokinetic measures

INTERVENTIONS:
Genetic: Blood drawn for genotyping — Blood will be drawn for genotyping (predefined list of genes) just before the start of sunitinib (baseline).
Biological: Blood drawn for pharmacokinetic measures — Blood will be drawn for pharmacokinetic measures between CmD15 and CmD28 of each sunitinib cycle.*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.

SUMMARY:
The primary objective of this study is to determine the percentage of patients with a plasma concentration of sunitinib remaining at equilibrium ([Suni]REq) greater than 100 ng / ml (effective concentration according to the current literature).

DETAILED DESCRIPTION:
The secondary objectives of this study are:

* To describe the distribution of constitutional genetic determinants related to sunitinib pharmacokinetics, and to study their correlation with

  * the [Suni]REq,
  * the advent of toxicity,
  * the tumor response.
* To describe the variation in the [Suni]REq and the plasma concentration of the active entity remaining at equilibrium ([ActEnt]REq) at:

  * the interindividual level,
  * overtime, between chemotherapy cycles.
* To describe the variation in the ratio of the plasma concentration of the metabolite remaining at equilibrium ([Metab]REq) to the [Suni]REq at:

  * the interindividual level,
  * overtime, between chemotherapy cycles.
* To explore potential correlations between the [Suni]REq and

  * toxicity,
  * tumor response.
* To explore potential correlations between the [ActEnt]REq and

  * toxicity,
  * tumor response.
* To explore potential correlations between the ratio [Metab]REq / [Suni]REq and

  * toxicity,
  * tumor response.

ELIGIBILITY:
Inclusion Criteria:

* The patient was correctly informed concerning the implementation of the study, its objectives, constraints and patient rights
* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient has kidney cancer and should begin treatment with sunitinib (Sutent) at the time of inclusion

Exclusion Criteria:

* The patient started treatment with sunitinib (Sutent) before inclusion
* The patient is participating in another interventional study
* The patient has participated in another interventional study within the last month
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication (or an incompatible drug combination) for a treatment used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with renal cell carcinoma treated with sunitinib (Sutent).
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with a plasma concentration of sunitinib remaining at equilibrium ([Suni]REq) greater than 100 ng / ml | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.

SECONDARY OUTCOMES:
Genotype: genetic polymorphisms of enzymes of phase I, phase II (conjugation), carriers of Phases 0 and III, the nuclear receptors PXR and CAR, pharmacological targets of sunitinib (tyrosine kinase receptors). | Baseline (day 0)
  Predefined list of genes:
  ABCB1 ABCC2 ABCG2 CYP1A1 CYP1A2 CYP2A6 CYP2B6 CYP2C19 CYP2C8 CYP2C9 CYP2D6 CYP2E1 CYP3A4 CYP3A5 NR1I2 NR1I3 SLC15A2 SLC22A1 SLC22A2 SLC22A6 SLCO1B1 SLCO1B3 SULT1A1 UGT1A1 UGT2B15 UGT2B17 UGT2B7 VEGFR1,2,3 PDGFR-α et β KIT
[Suni]REq per cure | Between CmD15* and CmD28* for 18 months
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
The presence/absence of grade I, II, III, IV, V (CTCAE version 4.0) toxicities per cure | 18 months
Tumor response per cure | 18 months
Toxicity (yes/no) for each type of toxic event per cure | Between CmD15* and CmD28* for 18 months
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
[Suni]REq at the 1st cure, averaged per initial dosing (37.5mg, 50 mg, 75 mg, 100mg) | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
the average [Suni]REq over all cures | 18 months
For each cure, the average [Suni]REq for cure 1 to cure m | 18 months
For each cure, the ratio of the plasma concentration of the metabolite remaining at equilibrium ([Metab]REq) / [Suni]REq | Between CmD15* and CmD28* for 18 months
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
[Metab]REq / [Suni]REq | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
[Metab]REq / [Suni]REq averaged per initial dosing | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
Mean [Metab]REq / [Suni]REq for all cures | 18 months
For each cure, the average [Metab]REq / [Suni]REq for cure 1 to cure m | 18 months
For each cure, the plasma concentration of the active entity remaining at equilibrium ([ActEnt]REq) | 18 months
[ActEnt]REq | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
[ActEnt]REq averaged per initial dosing | Between C1D15* and C1D28*
  *Each patient will undergo several cycles of treatment with sunitinib during the monitoring period as part of routine care (= 18 months; the number of cycles per patient can vary, which is normal). Each cycle and each day of the cycle will be annotated with the letters C and D, respectively, followed by a number in chronological order. Thus C1D1 refers to to the first day of the first cycle; CmDn will be the nth day of the mth cycle.
Mean [ActEnt]REq for all cures | 18 months
For each cure, the average [ActEnt]REq for cure 1 to cure m | 18 months
For each cure, the % of patients whose dosings were modified since the beginning of the study | 18 months
Presence/absence of side effects noted in the summary of product characteristics for sunitinib | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Litaty Mbatchi, PharmD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Institut de Cancérologie du Gard (ICG), Nîmes

REFERENCES:
- [Result] Mbatchi LC, Leenhardt F, Occean BV, Perrin O, Boyer JC, Gongora C, Pourquier P, Mura T, Chapelle A, Topart D, Evrard A, Houede N. Genetic polymorphisms of VEGFR2 and FGFR2 genes are associated with exposure to sunitinib and cardiovascular toxicity. Pharmacogenomics. 2025 Sep-Oct;26(13-14):485-493. doi: 10.1080/14622416.2025.2579001. Epub 2025 Nov 24. PMID 41277563